CLINICAL TRIAL: NCT05231811
Title: The Effect of Classical Foot Massage on Insomnia and an Anxiety in Preeclamptic Pregnant Women: A Randomized Controlled Study
Brief Title: Classic Foot Massage Applied to Preeclamptic Pregnants and Insomnia and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Collaborators: ayça şolt kırca (Unknown)
Responsible Party: Principal Investigator, NURDİLAN SENER, Asssistant professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: firat universityyyyy
Record Dates: First submitted 2022-01-26; First posted 2022-02-09 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Pregnant Women
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): During the massage; A pillow will be placed under the patient's leg and a disposable cover will be placed on the pillow. During the massage, pregnant women will be massaged with baby oil or vaseline cream. The soles of the pregnant women will be rubbed by the practitioner's fingers. The practitioner will make circular movements by applying pressure to the sole of the pregnant woman's feet with her thumb, and will apply pressure to the foot with up and down movements, using the joint protrusions on the upper surface of the hand that she has made into a fist. The heel and ankle will be squeezed between the thumb and forefinger of the researcher and kneaded and the massage will be terminated.
  Interventions: Other: massage
- control group (No Intervention): no intervention will be made in the control group

INTERVENTIONS:
Other: massage — Pregnant women by the researcher; Foot massage consisting of classical massage techniques will be applied in a room in the clinic reserved for this application. During the massage; A pillow will be placed under the patient's leg and a disposable cover will be placed on the pillow. During the massage, pregnant women will be massaged with baby oil or vaseline cream. The soles of the pregnant women will be rubbed by the practitioner's fingers. The practitioner will make circular movements by applying pressure to the sole of the pregnant woman's feet with her thumb, and will apply pressure to the foot with up and down movements, using the joint protrusions on the upper surface of the hand that she has made into a fist. The heel and ankle will be squeezed between the thumb and forefinger of the researcher and kneaded and the massage will be terminated. During the application, the researcher who performs the massage will pay attention to the precautions applied in the hospital.
  Arms: experimental group

SUMMARY:
Preeclampsia affects the sleep quality of pregnant women. With this study, it is expected that the sleep quality will be regulated by applying massage to pregnant women.

DETAILED DESCRIPTION:
One of the most important life events that cause change in a woman's life is the experience of pregnancy and childbirth. Pregnancy is a natural process for a woman; However, many women die due to complications during pregnancy. Severe hypertension is among the main causes of maternal and infant mortality during pregnancy and postpartum period. Hypertension in pregnancy occurs in 12-15% of all pregnancies, of which approximately 70% is preeclampsia and the remainder is chronic hypertension. It can cause severe hypertension, ablatio placenta, cerebral hemorrhage, pulmonary edema, liver and kidney failure, stroke, hemorrhage, intrauterine fetal death, HELLP (hemolysis, increased liver enzymes, low platelet) syndrome and maternal death in preeclamptic pregnant women. There is a relationship between hypertension and sleep disorders during pregnancy, . It has been reported that some sleep problems such as insomnia, fragmented sleep, snoring, sleep apnea and non-idiopathic insomnia are more common in pregnant women with preeclampsia than healthy pregnant women. Sleep disorders are associated with both increased morbidity and mortality. Poor sleep quality also increases the risk of depression. Sleep disorders also affect cardiovascular morbidity, including neuroendocrine, metabolic and inflammatory systems. Short sleep duration in pregnancy is also associated with longer delivery times and increased cesarean rates. Similarly, sleep problems experienced during pregnancy, poor sleep quality and stress may cause prolongation of labor, more fatigue of the mother during labor, development of complications, and increased fear and anxiety of the mother; It can lead to inadequate care of pregnant women, increase in the incidence of glucose intolerance and gestational diabetes, preterm delivery, delivery of a low-birth-weight baby and developmental problems in the baby. Moreover , it has been determined that the 3rd trimester sleep quality score is also associated with postpartum depressive symptoms . All these results show the importance of sleep for a healthy pregnancy. Various ways of coping are sought to solve sleep problems during pregnancy. These include lip exercises and diaphragmatic breathing exercises, training programs, yoga, passive exercises, and footbathing. In addition, it has been reported that applying foot massage to pregnant women with physiological edema in the lower extremities relieves insomnia complaints. It has been observed in the literature that classical foot massage performed in different disease groups reduces sleep symptoms. However, no study has been found in the literature examining the effect of classical foot massage applied to pregnant women with preeclampsia on insomnia. The aim of this study is to determine the effect of classical foot massage applied to preeclamptic pregnant women on sleep symptoms. If classical foot massage reduces insomnia symptoms, the effectiveness of a non-pharmacological method in reducing insomnia symptoms of preeclamptic pregnant women has been evaluated, and it is thought that a new approach will be presented both to the literature and to basic care interventions.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with preeclampsia
* Not having been diagnosed with pre-pregnancy sleep and not using one of the pharmacological or non-pharmacological treatment methods
* not using any medication for sleep

Exclusion Criteria:

* Having a history of psychiatric illness or receiving psychiatric treatment (Pharmacotherapy or psychotherapy) Pregnant women hospitalized for less than 1 week
* Having a chronic disease other than preeclampsia (Diabetes, Thyroid dysfunction, Cardio vascular problem, etc.)
* Pregnant women who lost their baby during the research period
* Obstetric or non-obstetric complications,
* Having any problem that prevents communication (such as not knowing Turkish, having a hearing, speaking and understanding disorder)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant woman
Enrollment: 71 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
The State Anxiety Inventory (STAI-2): | between 2 to 4 weeks
  The scale consists of twenty items and requires individuals to identify their feelings at a certain moment in particular situations and to answer the questions by considering how they feel about their current situation. Scores on the scale range between 20 and 80 1970. Öner and Le Compte (1974-1977) adapted the scale to Turkish culture and conducted its reliability and validity study [26]. The scale consists of twenty items and requires individuals to identify their feelings at a certain moment in particular situations and to answer the questions by considering how they feel about their current situation. Scores on the scale range between 20 and 80.

SECONDARY OUTCOMES:
The Insomnia Severity Index | betwee 2 to 4 weeks
  This seven-item scale was designed to identify the level of insomnia symptoms. It is utilized to screen the normal population and evaluate clinical insomnia [23-24]. Scores in the range of 0-4 are used to evaluate items on this 5-point Likerttype scale. Scores on the scale vary from 0 to 28, which are interpreted as follows: 0 to 7 refer to clinically insignificant insomnia; 8 to 14 refer to sub-threshold insomnia; 15 to 21 refer to moderate level of clinical insomnia; 22 to 28 refer to severe clinical insomnia

CONTACTS AND LOCATIONS:
Overall Officials: Nurdilan Şener, Principal Investigator — Firat University; AYÇA ŞOLT KIRCA, Study Director — Kırklareli University
Locations (2):
- Turkey (Türkiye) (2):
  - Ayça Şolt Kirca, Kırklareli, Kirklareli̇
  - NURDİLAN, Elâzığ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirca AS, Cetin NS. The effect of classical foot massage on insomnia and anxiety in preeclamptic pregnant women: a randomized controlled study. Rev Assoc Med Bras (1992). 2024 Feb 26;70(2):e20230744. doi: 10.1590/1806-9282.20230744. eCollection 2024. PMID 38422316